CLINICAL TRIAL: NCT02442765
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy, Safety, and Tolerability of AVP-786 (Deuterated [d6]-Dextromethorphan Hydrobromide [d6-DM]/Quinidine Sulfate [Q]) for the Treatment of Agitation in Patients With Dementia of the Alzheimer's Type
Brief Title: Efficacy, Safety and Tolerability of AVP-786 for the Treatment of Agitation in Patients With Dementia of the Alzheimer's Type
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-AVP-786-301
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Results first posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-01

CONDITIONS: Agitation in Patients With Dementia of the Alzheimer's Type
Keywords: Agitation; Dementia; Alzheimer's disease
MeSH Terms: conditions — Psychomotor Agitation; Dementia; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Sequential parallel comparison design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Stage 1: Placebo (Placebo Comparator): Participants received matching placebo orally twice daily (BID) for 6 weeks (Days 1-42) in Stage 1. Participants who completed Stage 1 were eligible to Participate in Stage 2.
  Interventions: Drug: Placebo
- Stage 1: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) (Experimental): Participants received AVP-786-18 mg orally once daily (QD) in the morning and placebo orally QD in the evening for the first 7 days, followed by AVP-786-18 mg orally BID for the remaining 5 weeks (Days 8-42). Participants who completed Stage 1 were eligible to participate in Stage 2.
  Interventions: Drug: AVP-786
- Stage 1: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg) (Experimental): Participants received AVP-786-18 mg orally QD in the morning and placebo orally QD in the evening for the first 7 days, followed by AVP-786-18 mg orally BID for 2 weeks (Days 8-21). From Day 22, participants received AVP-786-28 mg orally BID for the remaining 3 weeks. Participants who completed Stage 1 were eligible to participate in Stage 2.
  Interventions: Drug: AVP-786
- Stage 2: Placebo (Placebo Comparator): Participants who received matching placebo orally BID for 6 consecutive weeks in Stage 1 were re-randomized in Stage 2 to receive the study drug or placebo from Day 43 to Day 85.
  Interventions: Drug: Placebo
- Stage 1: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) to: Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) (Experimental): Participants who received AVP-786-18 mg in Stage 1 continued to receive AVP-786-18 mg orally BID for the 6 weeks (Days 43-85) in Stage 2..
  Interventions: Drug: AVP-786; Drug: Placebo
- Stage 1: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg) to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg) (Experimental): Participants who received AVP-786-28 mg in Stage 1 continued to receive AVP-786-28 mg orally BID for 6 weeks (Days 43-85) in Stage 2
  Interventions: Drug: AVP-786; Drug: Placebo
- Experimental: Stage 1: Placebo to: Stage 2: AVP-786-18 d6-DM 18 mg/Q 4.9 mg (Experimental): Participants who were placebo responders or non-responders in Stage 1 received AVP-786-18 for 1 week, orally, QD, followed by AVP-786-18 BID for 2 weeks; followed by AVP-786-28 BID for the last 3 weeks.
  Interventions: Drug: AVP-786; Drug: Placebo
- Stage 1: Placebo to: Stage 2: AVP-786-28 d6 DM 28 mg/Q 4.9 mg (Experimental): Participants who were placebo responders or non-responders in Stage 1 received AVP-786-28 for 1 week, orally, QD, followed by AVP-786-28 BID for 2 weeks; followed by AVP-786-28 BID for the last 3 weeks.
  Interventions: Drug: AVP-786; Drug: Placebo

INTERVENTIONS:
Drug: AVP-786
  Arms: Experimental: Stage 1: Placebo to: Stage 2: AVP-786-18 d6-DM 18 mg/Q 4.9 mg; Stage 1: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Stage 1: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) to: Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Stage 1: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Stage 1: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg) to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Stage 1: Placebo to: Stage 2: AVP-786-28 d6 DM 28 mg/Q 4.9 mg
Drug: Placebo
  Arms: Experimental: Stage 1: Placebo to: Stage 2: AVP-786-18 d6-DM 18 mg/Q 4.9 mg; Stage 1: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) to: Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Stage 1: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg) to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Stage 1: Placebo; Stage 1: Placebo to: Stage 2: AVP-786-28 d6 DM 28 mg/Q 4.9 mg; Stage 2: Placebo

SUMMARY:
Participants with agitation secondary to dementia of the Alzheimer's type. The diagnosis of probable Alzheimer's disease (AD) was to be based on the "2011 Diagnostic Guidelines for Alzheimer's Disease" issued by the National Institute on Aging (NIA)-Alzheimer's Association (AA) workgroups.

DETAILED DESCRIPTION:
Eligible participants for this study must have had a diagnosis of probable AD and must have had clinically meaningful agitation secondary to AD.

This was to be a multicenter, randomized, placebo-controlled study, consisting of 12 weeks of treatment.

Approximately 380 participants were to be enrolled at approximately 60 centers in North America.

Study medication was to be administered orally twice-daily from Day 1 through Day 85. Screening was to occur within approximately 4 weeks prior to randomization. Following screening procedures for assessment of inclusion and exclusion criteria, eligible participants were to be randomized into the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer's Disease (AD) according to the 2011 National Institute on Aging-Alzheimer's Association (NIA-AA) working groups criteria
* The participant has clinically significant, moderate/severe agitation at the time of screening and for at least 2 weeks prior to randomization
* The diagnosis of agitation must meet the International Psychogeriatric Association (IPA) provisional definition of agitation
* Either out patients or residents of an assisted-living facility or a skilled nursing home
* Clinical Global Impression of Severity of Illness (CGIS) score assessing Agitation is >= 4 (moderately ill) at screening and baseline
* Mini-Mental State Examination (MMSE) score is between 6 and 26 (inclusive) at screening and baseline
* Caregiver who is able and willing to comply with all required study procedures. In order to qualify as a reliable informant (i.e., caregiver) capable of assessing changes in participant's condition during the study, the individual must spend a minimum of 2 hours per day for 4 days per week with the participant.

Exclusion Criteria:

* Participant has dementia predominantly of non-Alzheimer's type (e.g., vascular dementia, frontotemporal dementia, Parkinson's disease, substance-induced dementia)
* Participants with co-existent clinically significant or unstable systemic diseases that could confound the interpretation of the safety results of the study (e.g., malignancy, poorly controlled diabetes, poorly controlled hypertension, unstable pulmonary, renal or hepatic disease, unstable ischemic cardiac disease, dilated cardiomyopathy, or unstable valvular heart disease)
* Participant with myasthenia gravis

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2015-07-23 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (106):
- United States (92):
  - Clinical Research Site, Phoenix, Arizona
  - Clinical Research Site, Scottsdale, Arizona
  - Clinical Research Site, Little Rock, Arkansas
  - Clinical Research Site#1, Irvine, California
  - Clinical Research Site#2, Irvine, California
  - Clinical Research Site, Long Beach, California
  - Clinical Research Site, Oceanside, California
  - Clinical Research Site, Orange, California
  - Clinical Research Site#1, San Diego, California
  - Clinical Research Site#2, San Diego, California
  - Clinical Research Site, Santa Ana, California
  - Clinical Research Site, Tustin, California
  - Clinical Research Site, Denver, Colorado
  - Clinical Research Site, Cromwell, Connecticut
  - Clinical Research Site, New London, Connecticut
  - Clinical Research Site, Norwalk, Connecticut
  - Clinical Research Site, Atlantis, Florida
  - Clinical Research Site, Boca Raton, Florida
  - Clinical Research Site, Brandon, Florida
  - Clinical Research Site#1, Coral Gables, Florida
  - Clinical Research Site#2, Coral Gables, Florida
  - Clinical Research Site#3, Coral Gables, Florida
  - Clinical Research Site#1, Deerfield Beach, Florida
  - Clinical Research Site, Doral, Florida
  - Clinical Research Site, Hialeah, Florida
  - Clinical Research Site#1, Hialeah, Florida
  - Clinical Research Site#2, Hialeah, Florida
  - Clinical Research Site, Jacksonville, Florida
  - Clinical Research Site, Kendall, Florida
  - Clinical Research Site, Kissimmee, Florida
  - Clinical Research Site, Lake Worth, Florida
  - Clinical Research Site, Miami, Florida
  - Clinical Research Site#1, Miami, Florida
  - Clinical Research Site#2, Miami, Florida
  - Clinical Research Site, Naples, Florida
  - Clinical Research Site, Oakland Park, Florida
  - Clinical Research Site, Orlando, Florida
  - Clinical Research Site, Ormond Beach, Florida
  - Clinical Research Site, Palm Beach Gardens, Florida
  - Clinical Research Site, Palmetto Bay, Florida
  - Clinical Research Site#2, Pompano Beach, Florida
  - Clinical Research Site, Sarasota, Florida
  - Clinical Research Site, St. Petersburg, Florida
  - Clinical Research Site#1, Tampa, Florida
  - Clinical Research Site#2, Tampa, Florida
  - Clinical Research Site, Tampa, Florida
  - Clinical Research Site, The Villages, Florida
  - Clinical Research Site, West Palm Beach, Florida
  - Clinical Research Site, Winter Park, Florida
  - Clinical Research Site, Atlanta, Georgia
  - Clinical Research Site, Newnan, Georgia
  - Clinical Research Site, Honolulu, Hawaii
  - Clinical Research Site, Schaumburg, Illinois
  - Clinical Research Site, Indianapolis, Indiana
  - Clinical Research Site, Lenexa, Kansas
  - Clinical Research Site, Paducah, Kentucky
  - Clinical Research Site, Bedford, Massachusetts
  - Clinical Research Site, Quincy, Massachusetts
  - Clinical Research Site, Ann Arbor, Michigan
  - Clinical Research Site, Paw Paw, Michigan
  - Clinical Research Site, Hattiesburg, Mississippi
  - Clinical Research Site, Creve Coeur, Missouri
  - Clinical Research Site, St Louis, Missouri
  - Clinical Research Site, Mount Arlington, New Jersey
  - Clinical Research Site, Toms River, New Jersey
  - Clinical Research Site, West Long Branch, New Jersey
  - Clinical Research Site, Amherst, New York
  - Clinical Research Site, Brooklyn, New York
  - Clinical Research Site, New York, New York
  - Clinical Research Site, Orangeburg, New York
  - Clinical Research Site, Rochester, New York
  - Clinical Research Site, Staten Island, New York
  - Clinical Research Site, Durham, North Carolina
  - Clinical Research Site, Winston-Salem, North Carolina
  - Clinical Research Site, Akron, Ohio
  - Clinical Research Site, Cincinnati, Ohio
  - Clinical Research Site#1, Columbus, Ohio
  - Clinical Research Site#2, Columbus, Ohio
  - Clinical Research Site, Dayton, Ohio
  - Clinical Research Site, Westerville, Ohio
  - Clinical Research Site, Edmond, Oklahoma
  - Clinical Research Site, Oklahoma City, Oklahoma
  - Clinical Research Site, Moosic, Pennsylvania
  - Clinical Research Site, Willow Grove, Pennsylvania
  - Clinical Research Site, East Providence, Rhode Island
  - Clinical Research Site, Charleston, South Carolina
  - Clinical Research Site#2, Cordova, Tennessee
  - Clinical Research Site, Dallas, Texas
  - Clinical Research Site, Irving, Texas
  - Clinical Research Site, Mansfield, Texas
  - Clinical Research Site, Clinton, Utah
  - Clinical Research Site, Woodstock, Vermont
- Estonia (3):
  - Clinical Research Site#1, Tallinn
  - Clinical Research Site#2, Tallinn
  - Clinical Research Site, Tartu
- Clinical Research Site, Mittweida, Germany
- Poland (7):
  - Clinical Research Site, Lublin, Lublin Voivodeship
  - Clinical Research Site, Bydgoszcz
  - Clinical Research Site, Kielce
  - Clinical Research Site, Lublin
  - Clinical Research Site, Poznan
  - Clinical Research Site, Pruszcz Gdański
  - Clinical Research Site, Siemianowice Śląskie
- Clinical Research Site, Torres Vedras, Portugal
- Puerto Rico (2):
  - Clinical Research Site, Bayamón
  - Clinical Research Site, San Juan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 695 participants were screened of these, 308 participants failed screening, 387 participants were randomized out of which 382 participants had at least 1 post baseline efficacy assessment. (Modified Intent-to-Treat { mITT} population).
Pre-assignment Details: This study was conducted in 2 stages. 387 participants were randomized to treatment in Stage 1 and all the participants completed Stage 1 and were re-randomized into Stage 2 to compare AVP-786 28 mg, AVP-786 18 mg and placebo in parallel group (PG) design. In Stage 2, participants randomized to active treatment in Stage 1 (AVP-786-18 or AVP-786-28) continued to receive the same treatment and those randomized to placebo in Stage 1 were re-randomized to AVP-786-18, AVP-786-28, or placebo.
Groups:
- Stage 1: Placebo to: Stage 2: AVP-786-28 d6-DM 18 mg/Q 4.9 mg: Participants who were placebo responders or non-responders in Stage 1 received AVP-786-18 for 1 week, orally, QD, followed by AVP-786-18 BID for 2 weeks; followed by AVP-786-28 BID for the last 3 weeks..
Period: Stage 1- (Days 1 to 42)
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg) | Stage 2: Placebo | Stage 1: Placebo to: Stage 2: AVP-786-28 d6-DM 18 mg/Q 4.9 mg | Stage 1: Placebo to: Stage 2: AVP-786-28 d6 DM 28 mg/Q 4.9 mg | Stage 1: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) to: Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg) to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg)
Started | 194 | 96 | 97 | 0 (For Stage 2, participants randomized to active treatment in Stage 1 (AVP-786-18 or AVP-786-28) continued to receive the same treatment and those randomized to placebo in Stage 1 were rerandomized to AVP-786-18, AVP-786-28, or placebo.) | 0 | 0 | 0 | 0
Completed | 194 | 96 | 97 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2- (Days 43 to 85)
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg) | Stage 2: Placebo | Stage 1: Placebo to: Stage 2: AVP-786-28 d6-DM 18 mg/Q 4.9 mg | Stage 1: Placebo to: Stage 2: AVP-786-28 d6 DM 28 mg/Q 4.9 mg | Stage 1: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) to: Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg) to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg)
Started | 0 | 0 | 0 | 63 (For Stage 2, participants randomized to active treatment in Stage 1 (AVP-786-18 or AVP-786-28) continued to receive the same treatment and those randomized to placebo in Stage 1 were rerandomized to AVP-786-18, AVP-786-28, or placebo.) | 96 | 97 | 65 | 66
Completed | 0 | 0 | 0 | 56 | 86 | 92 | 59 | 55
Not Completed | 0 | 0 | 0 | 7 | 10 | 5 | 6 | 11
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 6 | 1 | 1 | 5
Not completed — Death | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Study Participant Withdrawal by Parent or Guardian | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1
Not completed — Reason not specified | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data were collected in members of the Stage 1 Modified Intent-to-Treat (mITT) Population, comprised of all participants randomized in the study who had at least one post-Baseline efficacy assessment.
Groups:
- Placebo: In Stage 1, participants received matching placebo orally twice daily (BID).
- AVP-786-18: In Stage 1, participants received AVP-786-18 orally once daily (OD) in the morning and placebo orally OD in the evening for the first 7 days, followed by AVP-786-18 mg orally BID for the remaining 5 weeks. In Stage 2, participants continued to receive AVP-786-18 mg orally BID for 6 consecutive weeks.
- AVP-786-28: In Stage 1, participants received AVP-786-18 mg orally OD in the morning and placebo orally OD in the evening for the first 7 days, followed by AVP-786-18 mg orally BID for 2 weeks. From Day 22, participants received AVP-786-28 orally BID for the remaining 3 weeks. In Stage 2, participants continued to receive AVP-786-28 mg orally BID for 6 consecutive weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | AVP-786-18 | AVP-786-28 | Total
Number analyzed (Participants) | 191 | 94 | 97 | 382
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.6 (7.92) | 73.8 (8.39) | 74.6 (7.69) | 75.4 (8.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 47 | 54 | 213
  Male | 79 | 47 | 43 | 169
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 3 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 6 | 6 | 24
  White | 175 | 87 | 89 | 351
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Stage 1 and Stage 2: Change From Baseline in the Cohen-Mansfield Agitation Inventory (CMAI) Composite Score to Week 6 and Week 12
Description: The CMAI score is used to assess the frequency of manifestations of agitated behaviors in participants. The CMAI consists of 29 agitated behaviors that are rated on a 7-point scale of frequency: 1, never; 2, less than once a week; 3, once or twice a week; 4, several times a week; 5, once or twice a day; 6, several times a day; 7, several times an hour. The CMAI total score ranges from 29 to 203. Higher scores indicate worsening of the condition. Change from Baseline was calculated as the post-Baseline score minus the Baseline score.
Time Frame: Stage 1: Baseline, Week 6; Stage 2: Baseline (Week 6), Week 12
Population: Stage 1 Modified Intent-to-Treat (mITT) Population: all participants randomized in Stage 1 who had at least 1 post-Baseline efficacy assessment. Stage 2 mITT Population: all participants randomized in Stage 2 who had at least 1 efficacy assessment in Stage 2. Data were reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Stage 1: Placebo: Participants received a matching placebo orally twice daily (BID) for 6 weeks (Days 1-42) in Stage 1. Participants who completed Stage 1 were eligible to participate in Stage 2.
- Stage 1: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg): Participants received AVP-786-18 mg orally QD in the morning and placebo orally QD in the evening for the first 7 days, followed by AVP-786-18 mg orally BID for 2 weeks (Days 8-21). From Day 22, participants received AVP-786-28 mg orally BID for the remaining 3 weeks (Days 22-42). Participants who completed Stage 1 were eligible to participate in Stage 2.
- Stage 1: Placebo Non-responders to Stage 2: Placebo: Participants who received matching placebo in Stage 1 and were classified as non-responders (participants randomized to placebo in Stage 1 whose Clinical Global Impression of Severity of Illness scale for Agitation (CGIS-Agitation) score was ≤ 3 at Visit 4 (Day 43) and NPI- Agitation/Aggression Domain score has decreased by ≥ 25% from Baseline) were re-randomized to placebo and continued to receive placebo BID from Day 43 to Day 85 in Stage 2.
- Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg): Participants who received matching placebo in Stage 1 and were classified non-responders were re-randomized in Stage 2 to receive AVP-786-18 mg orally QD in the morning and placebo orally QD in the evening for the first 7 days of Stage 2 (Days 43-49), followed by AVP-786-18 mg orally BID for the remaining 5 weeks (Days 50-85).
- Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg): Participants who received matching placebo in Stage 1 and were classified non-responders were re-randomized in Stage 2 to receive AVP-786-18 mg orally QD in the morning and placebo orally QD in the evening for the first 7 days of Stage 2 (Days 43-49), followed by AVP-786-18 mg orally BID for 2 weeks (Days 50-63). From Day 64, participants received AVP-786-28 mg orally BID for the remaining 3 weeks (Days 64-85).
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg) | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg)
Number analyzed (Participants) | 188 | 92 | 97 | 40 | 40 | 44
units on a scale
  Stage 1 Baseline: number analyzed (Participants) | 188 | 92 | 97 | 0 | 0 | 0
  Stage 1 Baseline | 73.9 (22.23) | 72.3 (23.08) | 71.7 (23.57) |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 180 | 85 | 94 | 0 | 0 | 0
  Change from Baseline at Week 6 | -10.7 (15.29) | -13.9 (16.70) | -10.3 (13.54) |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 0 | 40 | 40 | 44
  Stage 2 Baseline |  |  |  | 66.0 (24.71) | 68.9 (20.79) | 65.3 (19.36)
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 0 | 40 | 40 | 44
  Change from Baseline at Week 12 |  |  |  | -1.6 (11.08) | -5.6 (11.78) | -4.9 (12.13)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.021, mixed model repeated measures (MMRM) — MMRMs include fixed effects of treatment, visit, treatment-by-visit, BL, BL-by-visit, and in the Stage 1 model, BL NPI AA, risk assessment for falls, BL concomitant antipsychotic medication use. Unstructured variance-covariance was used; Least Squares Mean Difference = -4.0, 95% CI 2-sided [-7.4 to -0.6]
Statistical Analysis 2: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.731, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.6, 95% CI 2-sided [-3.9 to 2.7]
Statistical Analysis 3: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.157, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -3.5, 95% CI 2-sided [-8.4 to 1.4]
Statistical Analysis 4: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.150, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -3.6, 95% CI 2-sided [-8.4 to 1.3]
Statistical Analysis 5: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.008, MMRM — [p-value comment as in outcome 1, analysis 1]; Sequential Parallel Comparison Design (SPCD) was used with weight = 0.6 for Stage 1 and 0.4 for Stage 2; MMRM weighted z-statistic = -2.65
Statistical Analysis 6: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg) vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.208, MMRM — [p-value comment as in outcome 1, analysis 1]; SPCD was used with weight = 0.6 for Stage 1 and 0.4 for Stage 2; MMRM weighted z-statistic = -1.26

2. Secondary Outcome: Least Squares Mean Modified Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (mADCS-CGIC)-Agitation Score at Week 6 and Week 12
Description: The intent of the ADCS version of the CGIC is to provide a means to reliably assess the global impression of change from Baseline in a clinical trial. The mADCS-CGIC is a modification of the ADCS-CGIC instrument that focuses specifically on agitation. The participants are asked to rate their impression of change from Baseline as: 1, marked improvement; 2, moderate improvement; 3, minimal improvement; 4, no change; 5, minimal worsening; 6, moderate worsening; 7, marked worsening. Baseline was defined as the last non-missing assessment prior to Stage 1 randomization. Treatment effects were estimated at each stage by analysis of covariance (ANCOVA) with fixed effects for treatment, Baseline CMAI Total score, and in the Stage 1 model, Baseline NPI AA (≤ 6 versus [vs] > 6), risk assessments for falls (normal/mild vs moderate/severe), Baseline concomitant use of antipsychotic medications (yes vs no). Missing values were imputed by last observation carried forward (LOCF) within each stage.
Time Frame: Stage 1 Week 6; Stage 2 Week 12
Population: Stage 1 and Stage 2 mITT Populations. Data were reported for only those participants contributing data to the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg: Participants received AVP-786-18 mg orally once daily (QD) in the morning and placebo orally QD in the evening for the first 7 days, followed by AVP-786-18 mg orally BID for the remaining 5 weeks (Days 8-42). Participants who completed Stage 1 were eligible to participate in Stage 2.
- Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg: Participants received AVP-786-18 mg orally QD in the morning and placebo orally QD in the evening for the first 7 days, followed by AVP-786-18 mg orally BID for 2 weeks (Days 8-21). From Day 22, participants received AVP-786-28 mg orally BID for the remaining 3 weeks (Days 22-42). Participants who completed Stage 1 were eligible to participate in Stage 2.
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg | Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg)
Number analyzed (Participants) | 184 | 90 | 96 | 40 | 40 | 42
score on a scale
  Stage 1 Week 6: number analyzed (Participants) | 184 | 90 | 96 | 0 | 0 | 0
  Stage 1 Week 6 | 3.4 (1.13) | 3.2 (1.24) | 3.3 (1.12) |  |  |
  Stage 2 Week 12: number analyzed (Participants) | 0 | 0 | 0 | 40 | 40 | 42
  Stage 2 Week 12 |  |  |  | 3.9 (0.18) | 3.3 (0.18) | 3.5 (0.17)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg; Test type: Superiority; p = 0.331, ANCOVA; Least Squares Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.1]
Statistical Analysis 2: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg; Test type: Superiority; p = 0.400, ANCOVA; Least Squares Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.2]
Statistical Analysis 3: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.014, ANCOVA; Least Squares Mean Difference = -0.6, 95% CI 2-sided [-1.1 to -0.1]
Statistical Analysis 4: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.145, ANCOVA; Least Squares Mean Difference = -0.4, 95% CI 2-sided [-0.9 to 0.1]
Statistical Analysis 5: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.012, ANCOVA; SPCD OLS weighted z-statistic = -2.51 — OLS = ordinary least squares
Statistical Analysis 6: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.097, ANCOVA; SPCD OLS weighted z-statistic = -1.66

3. Secondary Outcome: Stage 1 and Stage 2: Change From Baseline in the Neuropsychiatric Inventory (NPI) Agitation/Aggression Domain Score to Week 6 and Week 12
Description: The NPI is a retrospective interview covering 12 neuropsychiatric symptom domains and is used to evaluate psychopathology, neuropsychiatric manifestations, and caregiver distress. The Agitation/Aggression domain is designed to collect information on the behavioral aspects of agitation/aggression in participants with probable Alzheimer's Disease (AD) and clinically meaningful agitation secondary to AD. Each NPI domain is rated by the caregiver for symptom frequency and severity. Symptom frequency is rated as: 1, occasionally; 2, often; 3, frequently; 4, very frequently. Symptom severity is rated as: 1, mild; 2, moderate; 3, severe. The total domain score is calculated as the frequency score multiplied by the severity score and thus ranges from 1 to 12. Higher scores indicate worsening symptoms. Change from Baseline was calculated as the post-Baseline score minus the Baseline score.
Time Frame: Stage 1: Baseline, Week 6; Stage 2: Baseline (Week 6), Week 12
Population: Stage 1 and Stage 2 mITT Populations. Data were reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg | Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg)
Number analyzed (Participants) | 191 | 94 | 97 | 40 | 41 | 44
units on a scale
  Stage 1 Baseline: number analyzed (Participants) | 191 | 94 | 97 | 0 | 0 | 0
  Stage 1 Baseline | 7.1 (2.39) | 6.5 (1.94) | 7.2 (2.42) |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 183 | 87 | 94 | 0 | 0 | 0
  Change from Baseline at Week 6 | -1.8 (3.58) | -2.0 (3.03) | -2.1 (2.94) |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 0 | 40 | 41 | 44
  Stage 2 Baseline |  |  |  | 6.9 (2.84) | 6.3 (2.71) | 6.3 (2.81)
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 0 | 39 | 41 | 41
  Change from Baseline at Week 12 |  |  |  | -1.7 (3.00) | -0.8 (3.15) | -0.9 (3.35)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg; Test type: Superiority; p = 0.182, MMRM — [p-value comment as in outcome 1, analysis 1]; SPCD was used with weight = 0.6 for Stage 1 and 0.4 for Stage 2; Least Squares Mean Difference = -0.5, 95% CI 2-sided [-1.3 to 0.2]
Statistical Analysis 2: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg; Test type: Superiority; p = 0.390, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.3, 95% CI 2-sided [-1.1 to 0.4]
Statistical Analysis 3: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.462, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.5, 95% CI 2-sided [-0.8 to 1.7]
Statistical Analysis 4: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.528, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.4, 95% CI 2-sided [-0.8 to 1.6]
Statistical Analysis 5: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.695, ANCOVA — MMRMs include fixed effects of treatment, visit, treatment-by-visit, Baseline (BL), BL-by-visit, and in the Stage 1 model, BL NPI AA, risk assessment for falls, BL concomitant antipsychotic medication use. Unstructured variance-covariance was used; MMRM weighted z-statistic = -0.39
Statistical Analysis 6: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.904, ANCOVA — [p-value comment as in outcome 3, analysis 5]; MMRM weighted z-statistic = -0.12

4. Secondary Outcome: Stage 1 and Stage 2: Change From Baseline in the NPI Caregiver Distress Score to Week 6 and Week 12
Description: The NPI is a retrospective interview covering 12 neuropsychiatric symptom domains and is used to evaluate caregiver distress. Each NPI domain is rated by the caregiver for symptom frequency and severity. Symptom frequency is rated as: 1, occasionally; 2, often; 3, frequently; 4, very frequently. Symptom severity is rated as: 1, mild; 2, moderate; 3, marked severe. The total caregiver distress score is calculated as the frequency score multiplied by the severity score and thus ranges from 1 to 12. Higher scores indicate worsening symptoms. Change from Baseline was calculated as the post-Baseline score minus the Baseline score.
Time Frame: Stage 1: Baseline, Week 6; Stage 2: Baseline (Week 6), Week 12
Population: Stage 1 and Stage 2 mITT Populations. Data were reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg | Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg)
Number analyzed (Participants) | 164 | 77 | 85 | 39 | 38 | 43
units on a scale
  Stage 1 Baseline: number analyzed (Participants) | 164 | 77 | 85 | 0 | 0 | 0
  Stage 1 Baseline | 18.87 (9.026) | 18.90 (9.266) | 18.88 (10.015) |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 147 | 69 | 75 | 0 | 0 | 0
  Change from Baseline at Week 6 | -4.31 (7.979) | -5.48 (8.559) | -4.83 (7.736) |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 0 | 39 | 38 | 43
  Stage 2 Baseline |  |  |  | 17.33 (9.010) | 15.95 (7.241) | 16.89 (7.416)
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 0 | 37 | 33 | 36
  Change from Baseline at Week 12 |  |  |  | -0.73 (6.533) | -1.67 (5.666) | 0.44 (7.265)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg; Test type: Superiority; p = 0.247, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.2, 95% CI 2-sided [-3.2 to 0.8]
Statistical Analysis 2: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg; Test type: Superiority; p = 0.721, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.4, 95% CI 2-sided [-2.3 to 1.6]
Statistical Analysis 3: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.419, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.2, 95% CI 2-sided [-4.3 to 1.8]
Statistical Analysis 4: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.534, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.9, 95% CI 2-sided [-2.0 to 3.9]
Statistical Analysis 5: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.163, ANCOVA; MMRM weighted z-statistic = -1.40
Statistical Analysis 6: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.851, ANCOVA; MMRM weighted z-statistic = 0.19

5. Secondary Outcome: Stage 1 and Stage 2: Change From Baseline in the NPI Aberrant Motor Behavior Domain Score to Week 6 and Week 12
Description: The NPI is a retrospective interview covering 12 neuropsychiatric symptom domains and is used to evaluate aberrant motor behavior. Each NPI domain is rated by the caregiver for symptom frequency and severity. Symptom frequency is rated as: 1, occasionally; 2, often; 3, frequently; 4, very frequently. Symptom severity is rated as: 1, mild; 2, moderate; 3, severe. The total domain score is calculated as the frequency score multiplied by the severity score and thus ranges from 1 to 12. Higher scores indicate worsening of the symptoms. Change from Baseline was calculated as the post-Baseline score minus the Baseline score.
Time Frame: Stage 1: Baseline, Week 6; Stage 2: Baseline (Week 6), Week 12
Population: Stage 1 and Stage 2 mITT Populations. Data were reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg): Participants who received matching placebo in Stage 1 and were classified non-responders were re-randomized in Stage 2 to receive AVP-786-18 mg orally QD in the morning and placebo orally QD in the evening for the first 7 days of Stage 2 (Days 43-49), followed by AVP-786-18 mg orally BID for 2 weeks (Days 50-63). From Day 64, participants received AVP-786-28 mg orally BID for the remaining 3 weeks (Days 65-85).
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg | Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg)
Number analyzed (Participants) | 191 | 94 | 97 | 40 | 41 | 44
units on a scale
  Stage 1 Baseline: number analyzed (Participants) | 191 | 94 | 97 | 0 | 0 | 0
  Stage 1 Baseline | 5.1 (3.94) | 4.9 (3.77) | 5.1 (4.07) |  |  |
  Change from Baseline at Week 6 Stage 2 Baseline: number analyzed (Participants) | 183 | 87 | 94 | 0 | 0 | 0
  Change from Baseline at Week 6 Stage 2 Baseline | -0.9 (3.62) | -1.6 (3.74) | -0.7 (3.86) |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 0 | 40 | 41 | 44
  Stage 2 Baseline |  |  |  | 5.2 (3.79) | 4.0 (3.87) | 4.3 (4.32)
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 0 | 39 | 41 | 41
  Change from Baseline at Week 12 |  |  |  | -0.4 (2.16) | 0.6 (3.24) | 1.1 (3.54)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg; Test type: Superiority; p = 0.146, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.6, 95% CI 2-sided [-1.4 to 0.2]
Statistical Analysis 2: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg; Test type: Superiority; p = 0.399, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.3, 95% CI 2-sided [-0.4 to 1.1]
Statistical Analysis 3: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.283, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.7, 95% CI 2-sided [-0.6 to 2.0]
Statistical Analysis 4: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.065, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 1.2, 95% CI 2-sided [-0.1 to 2.5]
Statistical Analysis 5: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.829, ANCOVA; MMRM weighted z-statistic = -0.22
Statistical Analysis 6: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.052, ANCOVA; MMRM weighted z-statistic = 1.94

6. Secondary Outcome: Stage 1 and Stage 2: Change From Baseline in the Zarit Burden Interview (ZBI) Score to Week 6 and Week 12
Description: The ZBI is a 22-item scale used to assess the impact of a participant with dementia and also other illnesses on the caregiver's burden. For each item of the scale, the caregiver indicates how often they feel the burden (never, rarely, sometimes, quite frequently, or nearly always). The score ranges from 0 to 88 and is determined by adding the numbered responses of the individual items. Higher scores indicate greater caregiver distress. Change from Baseline was calculated as the post-Baseline score minus the Baseline score. Treatment effects were estimated at each stage by ANCOVA with fixed effects for treatment, Baseline, and in the Stage 1 model, Baseline NPI AA (≤ 6 versus > 6), risk assessments for falls (normal/mild versus moderate/severe), Baseline concomitant use of antipsychotic medications (yes versus no). Missing values were imputed by LOCF within each stage.
Time Frame: Stage 1: Baseline, Week 6; Stage 2: Baseline (Week 6), Week 12
Population: Stage 1 and Stage 2 mITT Populations. Overall number of participants analyzed are the number of participants with data available for analysis at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg | Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg)
Number analyzed (Participants) | 191 | 94 | 97 | 40 | 41 | 44
units on a scale
  Stage 1 Baseline: number analyzed (Participants) | 190 | 94 | 97 | 0 | 0 | 0
  Stage 1 Baseline | 30.9 (16.19) | 30.0 (16.96) | 33.0 (16.68) |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 190 | 94 | 97 | 0 | 0 | 0
  Change from Baseline at Week 6 | -1.4 (8.22) | -2.0 (8.44) | -2.7 (9.49) |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 0 | 40 | 41 | 44
  Stage 2 Baseline |  |  |  | 31.5 (15.24) | 32.0 (16.57) | 28.6 (16.76)
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 0 | 40 | 41 | 44
  Change from Baseline at Week 12 |  |  |  | -1.1 (7.65) | 1.4 (8.71) | -0.5 (7.05)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg; Test type: Superiority; p = 0.530, ANCOVA; Least Squares Mean Difference = -0.7, 95% CI 2-sided [-2.7 to 1.4]
Statistical Analysis 2: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg; Test type: Superiority; p = 0.326, ANCOVA; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-3.1 to 1.0]
Statistical Analysis 3: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.135, ANCOVA; Least Squares Mean Difference = 2.5, 95% CI 2-sided [-0.8 to 5.9]
Statistical Analysis 4: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.895, ANCOVA; Least Squares Mean Difference = 0.2, 95% CI 2-sided [-3.1 to 3.5]
Statistical Analysis 5: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.502, ANCOVA; SPCD OLS weighted Z-statistic = 0.67
Statistical Analysis 6: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.564, ANCOVA; SPCD OLS weighted Z-statistic = -0.58

7. Secondary Outcome: Stage 1 and Stage 2: Change From Baseline in the NPI Irritability/Lability Domain Score to Week 6 and Week 12
Description: The NPI is a retrospective interview covering 12 neuropsychiatric symptom domains, including the irritability/lability domain score. Each NPI domain is rated by the caregiver for symptom frequency and severity. Symptom frequency is rated as: 1, occasionally; 2, often; 3, frequently; 4, very frequently. Symptom severity is rated as: 1, mild; 2, moderate; 3, severe. The total domain score is calculated as the frequency score multiplied by the severity score and thus ranges from 1 to 12. Higher scores indicate worsening of the symptoms. Change from Baseline was calculated as the post-Baseline score minus the Baseline score.
Time Frame: Stage 1: Baseline, Week 6; Stage 2: Baseline (Week 6), Week 12
Population: Stage 1 and Stage 2: mITT Populations. Data were reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg | Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg)
Number analyzed (Participants) | 191 | 94 | 97 | 40 | 41 | 44
units on a scale
  Stage 1 Baseline: number analyzed (Participants) | 191 | 94 | 97 | 0 | 0 | 0
  Stage 1 Baseline | 5.1 (3.33) | 5.1 (3.62) | 5.2 (3.39) |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 183 | 87 | 94 | 0 | 0 | 0
  Change from Baseline at Week 6 | -1.1 (3.84) | -1.9 (3.71) | -1.4 (3.62) |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 0 | 40 | 41 | 44
  Stage 2 Baseline |  |  |  | 4.5 (3.99) | 5.3 (3.54) | 5.2 (3.64)
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 0 | 39 | 41 | 41
  Change from Baseline at Week 12 |  |  |  | 0.2 (3.19) | -1.3 (3.88) | -0.9 (3.45)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg; Test type: Superiority; p = 0.061, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.8, 95% CI 2-sided [-1.6 to 0.0]
Statistical Analysis 2: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg; Test type: Superiority; p = 0.400, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.3, 95% CI 2-sided [-1.1 to 0.5]
Statistical Analysis 3: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.115, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.1, 95% CI 2-sided [-2.4 to 0.3]
Statistical Analysis 4: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.264, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.8, 95% CI 2-sided [-2.1 to 0.6]
Statistical Analysis 5: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.015, ANCOVA; MMRM weighted z-statistic = -2.44
Statistical Analysis 6: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.163, ANCOVA; MMRM weighted z-statistic = -1.40

8. Secondary Outcome: Stage 1 and Stage 2: Change From Baseline in the NPI Total Score to Week 6 and Week 12
Description: NPI evaluates both frequency and severity of 12 neuropsychiatric disturbances including delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, motor disturbance, nighttime behaviors, as well as appetite/eating. Total domain score= frequency x severity and thus ranges from 1 to 12. NPI domain is rated by caregiver for symptom frequency and severity. Frequency is rated as: 1=occasionally, 2=often, 3= frequently, and 4=very frequently. Severity is rated as: 1=mild; 2= moderate, and 3=severe. Frequency and severity rating scales has defined anchor points to enhance reliability of caregiver responses. Caregiver distress is rated for each positive neuropsychiatric symptom using following anchored scores. It is rated as 0=not at all, 1=minimal, 3=moderate, 4=severe, 5=very severe. Total score is calculated by adding the individual Item scores, to yield a possible total scores of 0 to 144.
Time Frame: Stage 1: Baseline, Week 6; Stage 2: Baseline (Week 6), Week 12
Population: Stage 1 and Stage 2 mITT Populations. Data were reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg | Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg)
Number analyzed (Participants) | 191 | 94 | 97 | 40 | 41 | 44
units on a scale
  Stage 1 Baseline: number analyzed (Participants) | 191 | 94 | 97 | 0 | 0 | 0
  Stage 1 Baseline | 40.2 (17.95) | 39.4 (18.93) | 40.1 (19.98) |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 183 | 87 | 94 | 0 | 0 | 0
  Change from Baseline at Week 6 | -9.2 (17.41) | -13.2 (17.99) | -10.6 (16.09) |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 0 | 40 | 41 | 44
  Stage 2 Baseline |  |  |  | 39.2 (22.47) | 34.7 (14.16) | 34.6 (16.93)
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 0 | 39 | 41 | 41
  Change from Baseline at Week 12 |  |  |  | -5.1 (14.03) | -4.4 (12.92) | -0.1 (18.82)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg; Test type: Superiority; p = 0.050, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -3.9, 95% CI 2-sided [-7.8 to -0.0]
Statistical Analysis 2: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg; Test type: Superiority; p = 0.412, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.6, 95% CI 2-sided [-5.4 to 2.2]
Statistical Analysis 3: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.775, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-7.8 to 5.8]
Statistical Analysis 4: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.333, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 3.3, 95% CI 2-sided [-3.5 to 10.1]
Statistical Analysis 5: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.133, ANCOVA; MMRM weighted z-statistic = -1.50
Statistical Analysis 6: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.829, ANCOVA; MMRM weighted z-statistic = 0.22

9. Secondary Outcome: Stage 1 and Stage 2: Change From Baseline in the Clinical Global Impression of Severity of Illness (CGIS)-Agitation Domain Score to Week 6 and Week 12
Description: The CGIS-Agitation is an observer-rated scale that measures illness severity. CGIS is used to assess the severity of agitation. The CGIS score is rated on a 7-point scale (1 = normal, not at all ill; 7 = among the most extremely ill participants). Change from Baseline was calculated as the post-Baseline score minus the Baseline score. Treatment effects were estimated at each stage by ANCOVA with fixed effects for treatment, Baseline, and in the Stage 1 model, Baseline NPI AA (≤ 6 versus > 6), risk assessments for falls (normal/mild versus moderate/severe), Baseline concomitant use of antipsychotic medications (yes versus no). Missing values were imputed by LOCF within each stage.
Time Frame: Stage 1: Baseline, Week 6; Stage 2: Baseline (Week 6), Week 12
Population: Stage 1 and Stage 2 mITT Populations. Data were reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg | Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg)
Number analyzed (Participants) | 191 | 94 | 97 | 40 | 41 | 44
units on a scale
  Stage 1 Baseline: number analyzed (Participants) | 191 | 94 | 97 | 0 | 0 | 0
  Stage 1 Baseline | 4.5 (0.64) | 4.3 (0.49) | 4.4 (0.70) |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 191 | 94 | 97 | 0 | 0 | 0
  Change from Baseline at Week 6 | -0.5 (0.78) | -0.7 (0.97) | -0.7 (1.04) |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 0 | 40 | 41 | 44
  Stage 2 Baseline |  |  |  | 4.4 (0.87) | 4.2 (0.77) | 4.1 (0.77)
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 0 | 40 | 41 | 44
  Change from Baseline at Week 12 |  |  |  | -0.2 (0.58) | -0.4 (0.70) | -0.3 (1.01)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg; Test type: Superiority; p = 0.118, ANCOVA; Least Squares Mean Difference = -0.2, 95% CI 2-sided [-0.4 to 0.0]
Statistical Analysis 2: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg; Test type: Superiority; p = 0.191, ANCOVA; Least Squares Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.1]
Statistical Analysis 3: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.225, ANCOVA; Least Squares Mean Difference = -0.2, 95% CI 2-sided [-0.5 to 0.1]
Statistical Analysis 4: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.227, ANCOVA; Least Squares Mean Difference = -0.2, 95% CI 2-sided [-0.5 to 0.1]
Statistical Analysis 5: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.049, ANCOVA; SPCD OLS weighted z-statistic = -1.97
Statistical Analysis 6: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.075, ANCOVA; SPCD OLS weighted z-statistic = -1.78

10. Secondary Outcome: Stage 1 and Stage 2: Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (ADCS-CGIC) Rating at Week 6 and Week 12
Description: The ADCS-CGIC rating scale provides a reliable means to assess change from a Baseline level of global function within the time frame of the trial. ADCS-CGIC-Overall focuses on the clinician's observations of change in the participant's cognitive, functional, and behavioral performance. The ADCS-CGIC-Overall responses (1-7) are rated as: 1 = marked improvement, 2 = moderate improvement, 3 = minimal improvement, 4 = no change, 5 = minimal worsening, 6 = moderate worsening, or 7 = marked worsening. Treatment effects were estimated at each stage by ANCOVA with fixed effects for treatment, Baseline CMAI Total score, and in the Stage 1 model, Baseline NPI AA (≤ 6 versus > 6), risk assessments for falls (normal/mild versus moderate/severe), Baseline concomitant use of antipsychotic medications (yes versus no). Missing values were imputed by LOCF within each stage.
Time Frame: Stage 1: Baseline, Week 6; Stage 2: Baseline (Week 6), Week 12
Population: Stage 1 and Stage 2 mITT Populations. Data were reported for only those participants contributing data to the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg | Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg)
Number analyzed (Participants) | 183 | 90 | 96 | 40 | 40 | 42
units on a scale
  Stage 1 Week 6: number analyzed (Participants) | 183 | 90 | 96 | 0 | 0 | 0
  Stage 1 Week 6 | 3.7 (0.11) | 3.5 (0.14) | 3.6 (0.13) |  |  |
  Stage 2 Week 12: number analyzed (Participants) | 0 | 0 | 0 | 40 | 40 | 42
  Stage 2 Week 12 |  |  |  | 4.0 (0.17) | 3.6 (0.17) | 3.7 (0.16)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg; Test type: Superiority; p = 0.364, ANCOVA; Least Squares Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.1]
Statistical Analysis 2: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg; Test type: Superiority; p = 0.427, ANCOVA; Least Squares Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.2]
Statistical Analysis 3: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.098, ANCOVA; Least Squares Mean Difference = -0.4, 95% CI 2-sided [-0.9 to 0.1]
Statistical Analysis 4: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.168, ANCOVA; Least Squares Mean Difference = -0.3, 95% CI 2-sided [-0.8 to 0.1]
Statistical Analysis 5: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.063, ANCOVA; SPCD OLS weighted z-statistic = -1.86
Statistical Analysis 6: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.115, ANCOVA; SPCD OLS weighted z-statistic = -1.57

11. Secondary Outcome: Stage 1 and Stage 2: Patient Global Impression of Change (PGIC) Score at Week 6 and Week 12
Description: The PGIC is a 7-point (1-7) scale used to assess treatment response: 1 = very much improved, = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, or 7 = very much worse. Treatment effects were estimated at each stage by ANCOVA with fixed effects for treatment, Baseline CMAI Total score, and in the Stage 1 model, Baseline NPI AA (≤ 6 versus > 6), risk assessments for falls (normal/mild versus moderate/severe), Baseline concomitant use of antipsychotic medications (yes vs no). Missing values were imputed by LOCF within each stage.
Time Frame: Stage 1: Baseline, Week 6; Stage 2: Baseline (Week 6), Week 12
Population: Stage 1 and Stage 2 mITT Populations. Data were reported for only those participants contributing data to the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg | Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg)
Number analyzed (Participants) | 185 | 90 | 96 | 40 | 41 | 44
units on a scale
  Stage 1 Week 6: number analyzed (Participants) | 185 | 90 | 96 | 0 | 0 | 0
  Stage 1 Week 6 | 3.4 (0.12) | 3.0 (0.15) | 3.1 (0.14) |  |  |
  Stage 2 Week 12: number analyzed (Participants) | 0 | 0 | 0 | 40 | 41 | 44
  Stage 2 Week 12 |  |  |  | 3.6 (0.20) | 3.1 (0.20) | 3.3 (0.19)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg; Test type: Superiority; p = 0.014, ANCOVA; Least Squares Mean Difference = -0.4, 95% CI 2-sided [-0.6 to -0.1]
Statistical Analysis 2: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg; Test type: Superiority; p = 0.111, ANCOVA; Least Squares Mean Difference = -0.2, 95% CI 2-sided [-0.5 to 0.1]
Statistical Analysis 3: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.062, ANCOVA; Least Squares Mean Difference = -0.5, 95% CI 2-sided [-1.1 to 0.0]
Statistical Analysis 4: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.305, ANCOVA; Least Squares Mean Difference = -0.3, 95% CI 2-sided [-0.8 to 0.3]
Statistical Analysis 5: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.003, ANCOVA; SPCD OLS weighted z-statistic = -3.01
Statistical Analysis 6: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.073, ANCOVA; SPCD OLS weighted z-statistic = -1.79

12. Secondary Outcome: Stage 1 and Stage 2: Change From Baseline in the Dementia Quality of Life (DEMQOL) Score to Week 6 and Week 12
Description: The DEMQOL scale is used to evaluate health-related QOL in participants with dementia and their caregivers. There are 2 versions of the DEMQOL: a 28-item version (rated by the participant); and a 31-item version (DEMQOL-proxy, rated by the caregiver). Both versions are recommended for evaluating participants (and their caregivers) with mild to moderate dementia. The DEMQOL total score ranges from 28 to 112. The DEMQOL-proxy is used for participants with severe dementia; the total score ranges from 31 to 124. For both versions, higher scores indicate greater QOL. Change from Baseline was calculated as the post-Baseline score minus the Baseline score. Treatment effects were estimated at each stage by ANCOVA with fixed effects for treatment, Baseline, and in the Stage 1 model, Baseline NPI AA (≤ 6 vs > 6), risk assessments for falls (normal/mild vs moderate/severe), Baseline concomitant use of antipsychotic medications (yes vs no). Missing values were imputed by LOCF within each stage.
Time Frame: Stage 1: Baseline, Week 6; Stage 2: Baseline (Week 6), Week 12
Population: Stage 1 and Stage 2 mITT Populations. Data were reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg | Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg)
Number analyzed (Participants) | 133 | 69 | 72 | 24 | 30 | 32
units on a scale
  Stage 1 Baseline: number analyzed (Participants) | 133 | 69 | 72 | 0 | 0 | 0
  Stage 1 Baseline | 85.7 (10.63) | 82.9 (10.22) | 84.0 (11.98) |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 133 | 69 | 72 | 0 | 0 | 0
  Change from Baseline at Week 6 | 2.3 (8.26) | 3.5 (8.57) | 4.4 (10.79) |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 0 | 24 | 30 | 32
  Stage 2 Baseline |  |  |  | 86.8 (9.96) | 90.0 (9.51) | 87.8 (10.72)
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 0 | 24 | 30 | 32
  Change from Baseline at Week 12 |  |  |  | 2.5 (5.40) | 3.1 (9.52) | 1.1 (13.06)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg; Test type: Superiority; p = 0.909, ANCOVA; Least Squares Mean Difference = 0.1, 95% CI 2-sided [-2.2 to 2.5]
Statistical Analysis 2: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg; Test type: Superiority; p = 0.226, ANCOVA; Least Squares Mean Difference = 1.4, 95% CI 2-sided [-0.9 to 3.8]
Statistical Analysis 3: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.405, ANCOVA; Least Squares Mean Difference = 2.1, 95% CI 2-sided [-2.9 to 7.1]
Statistical Analysis 4: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.714, ANCOVA; Least Squares Mean Difference = -0.9, 95% CI 2-sided [-5.8 to 4.0]
Statistical Analysis 5: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.456, ANCOVA; SPCD OLS weighted z-statistic = 0.75
Statistical Analysis 6: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.678, ANCOVA; SPCD OLS weighted z-statistic = 0.42

13. Secondary Outcome: Stage 1 and Stage 2: Change From Baseline in the Cornell Scale for Depression in Dementia (CSDD) Score to Week 6 and Week 12
Description: The CSDD scale is used to assess signs/symptoms of major depression in participants with dementia. CSDD has 19 items, and each item is rated for severity on the following scale of 0 to 2 (0 =absent, 1= mild/intermittent 2=severe). CSDD score is calculated by summing non-missing scores from each item score. The scale ranges from 0-no depression to 38 maximum depressions. Scores above 10 indicate a probable major depression, above 18 indicate a definite major depression, and below 6 as a rule are associated with the absence of significant depressive symptoms. Higher score indicated maximum depression.
Time Frame: Stage 1: Baseline, Week 6; Stage 2: Baseline (Week 6), Week 12
Population: Stage 1 and Stage 2 mITT Populations. Data were reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg | Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg)
Number analyzed (Participants) | 191 | 94 | 97 | 40 | 41 | 44
units on a scale
  Stage 1 Baseline: number analyzed (Participants) | 191 | 94 | 97 | 0 | 0 | 0
  Stage 1 Baseline | 6.2 (2.24) | 6.3 (2.11) | 6.4 (2.19) |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 191 | 94 | 97 | 0 | 0 | 0
  Change from Baseline at Week 6 | -0.3 (3.01) | -0.7 (3.09) | -0.5 (2.93) |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 0 | 40 | 41 | 44
  Stage 2 Baseline |  |  |  | 6.6 (3.89) | 5.9 (2.78) | 6.8 (2.84)
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 0 | 40 | 41 | 44
  Change from Baseline at Week 12 |  |  |  | -0.4 (2.56) | -0.5 (2.36) | -0.3 (3.09)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg; Test type: Superiority; p = 0.278, ANCOVA; Least Squares Mean Difference = -0.4, 95% CI 2-sided [-1.1 to 0.3]
Statistical Analysis 2: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg; Test type: Superiority; p = 0.817, ANCOVA; Least Squares Mean Difference = -0.1, 95% CI 2-sided [-0.8 to 0.6]
Statistical Analysis 3: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.500, ANCOVA; Least Squares Mean Difference = -0.4, 95% CI 2-sided [-1.4 to 0.7]
Statistical Analysis 4: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.795, ANCOVA; Least Squares Mean Difference = 0.1, 95% CI 2-sided [-0.9 to 1.2]
Statistical Analysis 5: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.213, ANCOVA; SPCD OLS weighted z-statistic = -1.25
Statistical Analysis 6: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.985, ANCOVA; SPCD OLS weighted z-statistic = 0.02

14. Secondary Outcome: Stage 2: Percentage of Participants With General Medical Health Rating (GMHR) Score
Description: The GMHR is a global clinical rating for medical health, designed to quantify in a single number (1 to 4) the severity of general comorbidity in a participant with dementia. The ratings are: 1 = poor; 2 = fair; 3 = good; 4 = excellent to very good. Data was collected for the treatment arm groups as pre-specified in the protocol for this outcome measure.
Time Frame: Baseline; Week 12
Population: Stage 2 mITT population included all participants who were rerandomized in Stage 2 and had at least 1 efficacy assessment in Stage 2 (after Week 6). The data is reported for stage 2 only. Overall number analyzed are the number of participants with data available for analyses. The percentages are rounded off to the nearest whole number.
Measure: Number; unit: percentage of participants
Groups:
- Stage 1: Placebo to Stage 2: Placebo: Participants who received a matching placebo in Stage 1, continued to receive a matching placebo in Stage 2 for 6 weeks (Day 43 to Day 85).
- Stage 1: Placebo to: Stage 2: AVP-786-18 d6-DM 18 mg/Q 4.9 mg: Participants who were placebo responders or non-responders in Stage 1 received AVP-786-18 for 1 week, orally, QD, followed by AVP-786-18 BID for 2 weeks; followed by AVP-786-28 BID for the last 3 weeks.
- Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg to Stage 2: AVP-786-18 d6-DM 18 mg/Q 4.9 mg: Participants who received AVP-786-18 mg in Stage 1 continued to receive AVP-786-18 mg orally BID for the 6 weeks (Days 43-85) in Stage 2.
Arm/Group | Stage 1: Placebo to Stage 2: Placebo | Stage 1: Placebo to: Stage 2: AVP-786-18 d6-DM 18 mg/Q 4.9 mg | Stage 1: Placebo to: Stage 2: AVP-786-28 d6 DM 28 mg/Q 4.9 mg | Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg to Stage 2: AVP-786-18 d6-DM 18 mg/Q 4.9 mg | Stage 1: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg) to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg)
Number analyzed (Participants) | 62 | 64 | 65 | 94 | 97
percentage of participants
  Excellent to very good | 22.6 | 20.3 | 13.8 | 20.2 | 20.6
  Good | 59.7 | 64.1 | 58.5 | 58.5 | 62.9
  Fair | 11.3 | 7.8 | 16.9 | 13.8 | 11.3
  Poor | 0 | 0 | 0 | 0 | 0
  Missing | 6.5 | 7.8 | 10.8 | 7.4 | 5.2

15. Secondary Outcome: Stage 1 and Stage 2: Change From Baseline in the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) Score to Week 6 and Week 12
Description: The ADAS is designed to evaluate the cognitive and non-cognitive behavioral dysfunction characteristics of participants with AD. The cognitive subscale (ADAS-cog) consists of 11 subsets related to memory, praxis, and language. ADAS-cog scores range from 0 to 70. Higher scores indicate greater cognitive impairment. The ADAS-cog is assessed for participants with an Mini-Mental State Examination (MMSE) score of ≥10 at the Baseline Visit. Change from Baseline was calculated as the post-Baseline score minus the Baseline score. Treatment effects were estimated at each stage by ANCOVA with fixed effects for treatment, Baseline, and in the Stage 1 model, Baseline NPI AA (≤ 6 versus > 6), risk assessments for falls (normal/mild versus moderate/severe), Baseline concomitant use of antipsychotic medications (yes vs no). Missing values were imputed by LOCF within each stage.
Time Frame: Stage 1: Baseline, Week 6; Stage 2: Baseline (Week 6), Week 12
Population: Stage 1 and Stage 2 mITT Populations. Data were reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg | Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg)
Number analyzed (Participants) | 131 | 68 | 71 | 25 | 29 | 32
units on a scale
  Stage 1 Baseline: number analyzed (Participants) | 131 | 68 | 71 | 0 | 0 | 0
  Stage 1 Baseline | 25.8 (10.10) | 26.2 (8.99) | 25.3 (8.88) |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 130 | 68 | 71 | 0 | 0 | 0
  Change from Baseline at Week 6 | -0.5 (4.46) | -2.0 (4.28) | -0.5 (4.72) |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 0 | 25 | 27 | 32
  Stage 2 Baseline |  |  |  | 26.9 (9.56) | 27.0 (9.27) | 25.3 (10.91)
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 0 | 25 | 27 | 32
  Change from Baseline at Week 12 |  |  |  | -0.8 (5.05) | 0.3 (4.95) | 0.1 (5.47)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg; Test type: Superiority; p = 0.018, ANCOVA; Least Squares Mean Difference = -1.6, 95% CI 2-sided [-2.9 to -0.3]
Statistical Analysis 2: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg; Test type: Superiority; p = 0.956, ANCOVA; Least Squares Mean Difference = 0.0, 95% CI 2-sided [-1.3 to 1.3]
Statistical Analysis 3: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.451, ANCOVA; Least Squares Mean Difference = 1.1, 95% CI 2-sided [-1.8 to 4.0]
Statistical Analysis 4: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.519, ANCOVA; Least Squares Mean Difference = 0.9, 95% CI 2-sided [-1.9 to 3.7]
Statistical Analysis 5: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg); Test type: Superiority; p = 0.471, ANCOVA; SPCD OLS weighted z-statistic = -0.72
Statistical Analysis 6: Comparison: Stage 1: Placebo vs Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg vs Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg); Test type: Superiority; p = 0.618, ANCOVA; SPCD OLS weighted z-statistic = 0.50

16. Secondary Outcome: Stage 1: Resource Utilization in Dementia (RUD): Percentage of Caregiver Who Reported That Their Responsibilities Affected Their Work and Who Visited Health Care Professionals
Description: RUD evaluates dementia participants utilization of formal and informal healthcare resources, including hospitalizations and doctor visits, living assistance, and time spent by nonprofessional caregivers. The RUD is administered as a semi-structured interview with the participant's primary caregiver and contains 2 sections; one focusing on caregiver impact (loss of work and leisure time incurred by caregiver) and the other focusing on the participant's use of healthcare resources. Information of caregivers who reported their responsibilities affected their work and who visited healthcare professionals from the interviews during Stage 1 is reported for this outcome measure. Data was collected for the treatment arm groups as pre-specified in the protocol for this outcome measure.
Time Frame: Stage 1: Week 6
Population: Stage 1 mITT Populations. Data were reported for only those participants contributing data to the analysis. Number analyzed are the number of participants available at the given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg)
Number analyzed (Participants) | 191 | 94 | 97
percentage of participants
  Caregivers Who Reported that their Responsibilities Affected Their Work: number analyzed (Participants) | 74 | 35 | 38
  Caregivers Who Reported that their Responsibilities Affected Their Work | 33.8 | 22.9 | 34.2
  Caregivers Who Visited Health Care Professionals: number analyzed (Participants) | 185 | 90 | 96
  Caregivers Who Visited Health Care Professionals | 42.2 | 31.1 | 44.8

17. Secondary Outcome: Stage 2: Resource Utilization in Dementia (RUD): Percentage of Caregiver Who Reported That Their Responsibilities Affected Their Work and Who Visited Health Care Professionals
Description: RUD evaluates dementia participants utilization of formal and informal healthcare resources, including hospitalizations and doctor visits, living assistance, and time spent by nonprofessional caregivers. The RUD is administered as a semi-structured interview with the participant's primary caregiver and contains 2 sections; one focusing on caregiver impact (loss of work and leisure time incurred by caregiver) and the other focusing on the participant's use of healthcare resources. Information of caregivers who reported their responsibilities affected their work and who visited healthcare professionals from the interviews during Stage 2 is reported for this outcome measure. Data was collected for the treatment arm groups as pre-specified in the protocol for this outcome measure.
Time Frame: Stage 2: Week 12
Population: Stage 2 mITT Population. Data were reported for only those participants contributing data to the analysis. Number analyzed are the number of participants available at the given timepoint.
Measure: Number; unit: percentage of participants
Groups:
- Stage 2: Placebo/Placebo: Participants who received matching placebo orally BID for 6 consecutive weeks in Stage 1 were re-randomized in Stage 2 to receive the study drug or placebo from Day 43 to Day 85.
Arm/Group | Stage 2: Placebo/Placebo | Stage 1: Placebo to: Stage 2: AVP-786-18 d6-DM 18 mg/Q 4.9 mg | Stage 1: Placebo to: Stage 2: AVP-786-28 d6 DM 28 mg/Q 4.9 mg | Stage 1: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) to: Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg) to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg)
Number analyzed (Participants) | 62 | 59 | 60 | 94 | 97
percentage of participants
  Caregivers Who Reported that their Responsibilities Affected Their Work: number analyzed (Participants) | 25 | 59 | 60 | 33 | 34
  Caregivers Who Reported that their Responsibilities Affected Their Work | 44.0 | 28.6 | 36.4 | 24.2 | 35.3
  Caregivers Who Visited Health Care Professionals: number analyzed (Participants) | 58 | 59 | 58 | 86 | 92
  Caregivers Who Visited Health Care Professionals | 43.1 | 30.5 | 29.3 | 26.7 | 37.0

18. Secondary Outcome: Stage 1: Resource Utilization in Dementia (RUD): Number of Hours Per Day the Caregiver Spent Assisting the Participant
Description: RUD evaluates dementia participants utilization of formal, informal healthcare resources, including hospitalizations, doctor visits, living assistance, time spent by nonprofessional caregivers. Information on hours per day caregiver spent assisting participant from interviews during Stage 1 is reported for this outcome measure, where the following questions (Q), Q1= On typical care day during last 30 days, how much time per day did you assist participant with tasks such as toilet visits, eating, dressing, grooming, walking, bathing? Q2= On typical care day during the last 30 days, how much time per day did you assist participant with tasks as (shopping, food preparation, housekeeping, laundry, transportation, taking medication, managing financial matters?; Q3= On typical care day during last 30 days, how much time per day did you spend supervising (preventing dangerous events)?(Q3). Data is collected for treatment arm groups as pre-specified in protocol for this outcome measure.
Time Frame: Stage 1: Week 6
Population: Stage 1 mITT Populations. Data were reported for only those participants contributing data to the analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg)
Number analyzed (Participants) | 171 | 84 | 90
hours
  Week 6 (Q1) | 2.0 [0 to 20] | 2.0 [0 to 24] | 2.0 [0 to 15]
  Week 6 (Q2) | 4.0 [1 to 24] | 4.0 [0 to 18] | 4.0 [1 to 15]
  Week 6 (Q3) | 3.0 [0 to 24] | 2.0 [0 to 24] | 2.8 [0 to 24]

19. Secondary Outcome: Stage 2: Resource Utilization in Dementia (RUD): Number of Hours Per Day the Caregiver Spent Assisting the Participant
Description: as for outcome 18
Time Frame: Stage 2: Week 12
Population: Stage 2 mITT Population. The data is reported for stage 2 only. Data were reported for only those participants contributing data to the analysis
Measure: Median (Full Range); unit: hours
Groups:
- Stage 1: Placebo to Stage 2: Placebo: Participants who received matching placebo in Stage 1, continued to receive matching placebo in Stage 2 for 6 weeks (Day 43 to Day 85).
- Stage 1: Placebo to Stage 2: AVP-786 18 mg: Participants who received matching placebo in Stage 1 were re-randomized to AVP-786-18 mg and received AVP-786-18 mg orally QD in the morning and placebo orally QD in the evening for the first 7 days of Stage 2 (Days 43-49), followed by AVP-786-18 mg orally BID for the remaining 5 weeks (Days 50-85).
- Stage 1: Placebo to Stage 2: AVP-786 28 mg: Participants who received matching placebo in Stage 1 were re-randomized to AVP-786-28 mg and received AVP-786-18 mg orally QD in the morning and placebo orally QD in the evening for the first 7 days of Stage 2 (Days 43-49), followed by AVP-786-18 mg orally BID for 2 weeks (Days 50-63). From Day 64, participants received AVP-786-28 mg orally BID for the remaining 3 weeks (Days 64-85).
Arm/Group | Stage 1: Placebo to Stage 2: Placebo | Stage 1: Placebo to Stage 2: AVP-786 18 mg | Stage 1: Placebo to Stage 2: AVP-786 28 mg | Stage 1: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) to: Stage 2: AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) | Stage 1: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg) to Stage 2: AVP-786-28 (d6-DM 28 mg/Q 4.9 mg)
Number analyzed (Participants) | 54 | 55 | 53 | 81 | 87
hours
  Week 12 (Q1) | 1.5 [0 to 15] | 2.0 [0 to 7] | 2.0 [0 to 12] | 2.0 [0 to 10] | 2.0 [0 to 14]
  Week 12 (Q2) | 4.0 [0 to 16] | 4.0 [0 to 24] | 4.0 [0 to 24] | 4.0 [0 to 17] | 4.0 [0 to 15]
  Week 12 (Q3) | 1.0 [0 to 19] | 3.0 [0 to 24] | 3.0 [0 to 20] | 2.0 [0 to 24] | 2.0 [0 to 18]

20. Secondary Outcome: Stage 1: Resource Utilization in Dementia (RUD) Score: Number of Days the Caregiver Spent Assisting the Participant
Description: RUD evaluates dementia participants utilization of formal, informal healthcare resources, including hospitalizations, doctor visits, living assistance, time spent by nonprofessional caregivers. Information on days caregiver spent assisting participant from interviews during Stage 1 is reported for outcome measure, where following questions (Q), Q1= During last 30 days, how many days did you spend providing these (toilet visits, eating, dressing, grooming, walking, bathing) services to participant?; Q2= On typical care day during last 30 days, how much time per day did you assist participant with tasks such as shopping, food preparation, housekeeping, laundry, transportation, taking medication, managing financial matters?; Q3= During last 30 days, how many days did you spend providing these services (supervising) to the participant?. Data is collected for the treatment arm groups as pre-specified in the protocol for this outcome measure.
Time Frame: Stage 1: Week 6
Population: Stage 1 mITT Populations. Data were reported for only those participants contributing data to the analysis.
Measure: Median (Full Range); unit: days
Groups:
- Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg: Participants received AVP-786-18 mg orally QD in the morning and placebo orally QD in the evening for the first 7 days, followed by AVP-786-18 mg orally BID for 2 weeks (Days 8-21). From Day 22, participants received AVP-786-28 mg orally BID for the remaining 3 weeks. Participants who completed Stage 1 were eligible to participate in Stage 2.
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786-18 d6-DM 18 mg/Q 4.9 mg | Stage 1: AVP-786-28 d6-DM 28 mg/Q 4.9 mg
Number analyzed (Participants) | 191 | 94 | 97
days
  Week 6 (Q1): number analyzed (Participants) | 171 | 84 | 90
  Week 6 (Q1) | 30.0 [0 to 30] | 30.0 [0 to 30] | 30.0 [0 to 30]
  Week 6 (Q2): number analyzed (Participants) | 171 | 84 | 90
  Week 6 (Q2) | 30.0 [0 to 30] | 30.0 [0 to 39] | 30.0 [4 to 30]
  Week 6 (Q3): number analyzed (Participants) | 171 | 84 | 90
  Week 6 (Q3) | 30.0 [0 to 30] | 30.0 [0 to 30] | 30.0 [0 to 30]

21. Secondary Outcome: 12-Week Parallel Group: Resource Utilization in Dementia (RUD) Score: Number of Days the Caregiver Spent Assisting the Participant
Description: as for outcome 20
Time Frame: 12-Week Parallel Group: Week 12
Population: mITT 12-Week Parallel-Group Population included all participants in the 12-Week Parallel Group who have at least one post-baseline efficacy assessment
Measure: Median (Full Range); unit: days
Arm/Group | Stage 1: Placebo to Stage 2: Placebo | Stage 1: Placebo to Stage 2: AVP-786 18 mg | Stage 1: Placebo to Stage 2: AVP-786 28 mg
Number analyzed (Participants) | 62 | 94 | 97
days
  Week 12 (Q1): number analyzed (Participants) | 54 | 81 | 87
  Week 12 (Q1) | 30.0 [0 to 30] | 30.0 [0 to 30] | 30.0 [0 to 30]
  Week 12 (Q2): number analyzed (Participants) | 54 | 81 | 87
  Week 12 (Q2) | 30.0 [0 to 30] | 30.0 [0 to 30] | 30.0 [0 to 30]
  Week 12 (Q3): number analyzed (Participants) | 54 | 81 | 87
  Week 12 (Q3) | 30.0 [0 to 30] | 30.0 [0 to 30] | 30.0 [0 to 30]

ADVERSE EVENTS:
Time Frame: Start of treatment up to Week 16 (End of treatment plus 30 days)
Description: Treatment-emergent adverse events (TEAEs), defined as those adverse events that began or worsened on or after the first dose date and before the last dose date + 30 days, are reported. TEAEs were collected in members of the Safety Population, comprised of all randomized participants who received at least one dose of study treatment.Safety data were summarized based on the treatment the participants received at any time during the study.
Groups:
- Placebo: Participants received a matching placebo orally twice daily (BID) for 6 weeks (Days 1-42) in Stage 1. Participants who completed Stage 1 were eligible to participate in Stage 2.
- AVP-786-18: Participants received AVP-786-18 mg orally once daily (QD) in the morning and placebo orally QD in the evening for the first 7 days, followed by AVP-786-18 mg orally BID for the remaining 5 weeks (Days 8-42). Participants who completed Stage 1 were eligible to participate in Stage 2.
- AVP-786-28: Participants received AVP-786-18 mg orally QD in the morning and placebo orally QD in the evening for the first 7 days, followed by AVP-786-18 mg orally BID for 2 weeks (Days 8-21). From Day 22, participants received AVP-786-28 mg orally BID for the remaining 3 weeks (Days 22-42). Participants who completed Stage 1 were eligible to participate in Stage 2.
Arm/Group | Placebo | AVP-786-18 | AVP-786-28
All-Cause Mortality (participants affected / at risk) | 1/194 | 3/156 | 1/159
Serious Adverse Events (participants affected / at risk) | 6/194 | 17/156 | 7/159
Other Adverse Events (participants affected / at risk) | 84/194 | 78/156 | 71/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=194) | AVP-786-18 (N=156) | AVP-786-28 (N=159)
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Injury associated with device (General disorders) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Hydroureter (Renal and urinary disorders) | 0 | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=194) | AVP-786-18 (N=156) | AVP-786-28 (N=159)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 4 | 2
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 2
Bundle branch block left (Cardiac disorders) | 0 | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Type V hyperlipidaemia (Congenital, familial and genetic disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 1
Eye allergy (Eye disorders) | 0 | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 10 | 7
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 4 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Poor dental condition (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 4 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 3 | 1 | 2
Feeling cold (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 3 | 0
Gait disturbance (General disorders) | 1 | 2 | 0
Asthenia (General disorders) | 0 | 1 | 0
Pain (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 9 | 9 | 5
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 3
Nasopharyngitis (Infections and infestations) | 3 | 0 | 3
Cellulitis (Infections and infestations) | 0 | 1 | 2
Fungal infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 2 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
Arthritis infective (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0
Helicobacter infection (Infections and infestations) | 1 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 12 | 14 | 12
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 4 | 5 | 2
Laceration (Injury, poisoning and procedural complications) | 0 | 3 | 1
Animal scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Conjunctival laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 3 | 3
Neutrophil count increased (Investigations) | 0 | 1 | 2
White blood cell count increased (Investigations) | 0 | 2 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 1
White blood cells urine positive (Investigations) | 0 | 0 | 1
Blood urea increased (Investigations) | 1 | 2 | 0
Electrocardiogram ST segment depression (Investigations) | 0 | 2 | 0
Weight increased (Investigations) | 1 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Blood glucose increased (Investigations) | 1 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0
Crystal urine (Investigations) | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1 | 0
Fungal test positive (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Glucose urine present (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0
Lymphocyte count increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Dizziness (Nervous system disorders) | 5 | 5 | 5
Somnolence (Nervous system disorders) | 7 | 6 | 4
Headache (Nervous system disorders) | 3 | 10 | 2
Lethargy (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 1 | 1 | 1
Decreased vibratory sense (Nervous system disorders) | 0 | 0 | 1
Hyperreflexia (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 2 | 0
Dyskinesia (Nervous system disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 10 | 4 | 7
Hallucination (Psychiatric disorders) | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 0 | 2
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 1
Hypnopompic hallucination (Psychiatric disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 4 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Glycosuria (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Spontaneous penile erection (Reproductive system and breast disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pemphigus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 2 | 2
Hot flush (Vascular disorders) | 0 | 1 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-05-16): https://cdn.clinicaltrials.gov/large-docs/65/NCT02442765/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/65/NCT02442765/SAP_001.pdf